CLINICAL TRIAL: NCT03843346
Title: The Impact of the 21 Gene Recurrence Score (RS) on Chemotherapy Prescribing in Estrogen Receptor Positive, Lymph Node Positive Early Stage Breast Cancer in Ireland
Brief Title: The Impact of the Gene Recurrence Score on Chemotherapy Prescribing in ER Positive, Lymph Node Positive Early Stage Breast Cancer
Status: Completed | Type: Observational
Sponsor: Cancer Trials Ireland (Network)
Responsible Party: Sponsor
Other Study IDs: CTRIAL-IE 15-34
Record Dates: First submitted 2018-10-11; First posted 2019-02-18 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue will be sent for 21 gene RS (OncotypeDx(r)) testing to Genomic Health as per standard clinical practice for patients with node negative tumours.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Postoperative group: Consists of 75 patients who have completed definite surgery for their primary breast cancer as determined by a Consultant Surgeon and have been referred to a Medical Oncologist for consideration of adjuvant chemotherapy.
  * Tumours of any size will be eligible
  * Between 1 and 3 lymph nodes involved by tumour as assessed by Consultant Pathologist
  * Micro metastases (<=0.2mm) will be eligibile
  * Isolated tumour cells only (node negative i+/i-) are excluded
- Cohort 2: Preoperative group: Consists of 75 patients who have been referred by a Consultant Surgeon to a Medical Oncologist for consideration of neoadjuvant (preoperative) chemotherapy.
  * Min tumour size 2.1mm (T2)
  * Histological proof of involvement of at 1 lymph node, including micrometastases (<=0.2mm)

SUMMARY:
This study examines the impact of an additional tumour test called the 21 gene Recurrence Score (OncotypeDx®), a commercially available test on a Medical Oncologist's decision to recommend chemotherapy.

DETAILED DESCRIPTION:
After a breast cancer and any lymph glands have been surgically removed, further (adjuvant) treatment is generally given to reduce the risk of cancer recurrence. For patients with estrogen receptor (ER) positive breast cancer, this treatment has traditionally been chemotherapy and hormone therapy. However, it is increasingly recognised that tumours which are ER positive and negative for the human epidermal growth factor receptor 2 (HER2), are relatively resistant to chemotherapy. It is likely that many more people are exposed to the risks for chemotherapy than ever benefit from it. In order to select patients who will get more benefit from chemotherapy and to spare those who get very little benefit from side effects, risk assessment tools are being developed.

The 21 Gene Recurrence Score is a test that examines the tumour genes to estimate the risk of the tumour relapsing and possible chemotherapy benefits. Currently, the 21 Gene Recurrence Score (OncotypeDx®) is used In Ireland for patients with no cancer in their lymph nodes. For these patients it can help in deciding who should get chemotherapy. Patients with low scores can sometimes avoid chemotherapy. In some countries, this test is offered to almost all patients with ER positive breast cancer, irrespective of whether the cancer has spread to lymph nodes or not. However, in Ireland this test is not standardly available for patients who have breast cancer involving lymph nodes.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria (All Patients)

1. Age 18 years of age or older
2. ER Positive Tumours (≥1% positive cells or Allred score ≥ 2 (Appendix 1))
3. Human Epidermal Growth Factor Receptor 2 (HER2) negative breast cancer (0-1 by IHC or FISH <2.0)
4. No evidence of metastatic disease on CT, bone scan or other imaging
5. Fit for consideration of chemotherapy as determined by the Investigator
6. Adequate performance status (Eastern Cooperative Oncology Group (ECOG) 0 or 1 (Appendix 2))

Inclusion Criteria - Cohort 1 (Postoperative Patients): N= 75

1. Adequate surgical excision of breast tumour (mastectomy or lumpectomy) and lymph nodes (sentinel lymph biopsy or axillary dissection)
2. Any tumour size (T stage (Appendix 3))
3. Involvement of 1-3 lymph nodes (N1, including micrometastases)

Inclusion Criteria - Cohort 2 (Preoperative Patients): N= 75

1. Candidates for preoperative therapy for early breast cancer
2. T2-T4 tumours
3. Involvement of at least one lymph node, (including micrometastases) on biopsy
4. Adequate tissue from core biopsy for 21 gene RS testing (approximate minimum 5mm)

Exclusion Criteria (All patients):

1. ER negative tumour (Allred score 0-1)
2. HER2 positive tumours as defined by IHC 3+ or FISH ≥ 2.0
3. Node negative disease, including those with Isolated tumour cells only (node negative i+/i-)
4. Known metastatic breast cancer
5. Performance status ≥ 2
6. Patients not considered by their treating physician to be fit to undergo chemotherapy.
7. Men with breast cancer.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The study will examine 2 cohorts of patients;
  * 75 patients (cohort 1; "postoperative") who have undergone resection of their primary breast cancer and
  * 75 patients (cohort 2; "preoperative") who are referred to a Medical Oncologist for consideration of neoadjuvant (preoperative) treatment.
  Both cohorts will have ER positive, lymph node positive breast cancer and both cohorts will undergo testing with the 21 gene RS.
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2017-03-16 (Actual); Primary Completion 2021-02-02 (Actual); Study Completion 2021-02-02 (Actual)

PRIMARY OUTCOMES:
Recommended Chemotherapy | 3 years
  The percentage reduction in the number of patients for whom chemotherapy is recommended following resection of their primary breast cancer and testing with the 21 gene RS (cohort 1; n=75)

SECONDARY OUTCOMES:
Impact of gene RS | 3 years
  Examine the impact of the 21 gene RS on chemotherapy recommendations in operable breast cancer in the postoperative and preoperative setting (cohorts 1 and 2; n=150) using questionnaires completed by Medical Oncologists.
Complete Response | 3 years
  Investigate the correlation between the 21 gene RS and pathological complete response from preoperative therapy in operable breast cancer (cohort 2; n=75).
Radiological Response Rate | 3 years
  Determine whether the 21 gene RS correlates with clinical, radiological response rate and the MD Anderson residual cancer burden score following preoperative therapy (cohort 2; n=75).
Economic Impact | 3 years
  Determine the economic impact of the 21 gene RS testing on ER positive, node positive breast cancer patients (cohorts 1 and 2; n=150) using a simple budget impact model

CONTACTS AND LOCATIONS:
Overall Officials: Dr Patrick Morris, Principal Investigator — Beaumont Hospital
Locations (10):
- Ireland (10):
  - Letterkenny University Hospital, Letterkenny, Co. Donegal
  - St Vincent's University Hospital, Dublin, Dublin 4
  - Mater Misericordiae University Hospital & Mater Private Hospital, Dublin, Dublin 7
  - Beaumont Hospital, Dublin, Dublin 9
  - Bon Secour Cork, Cork
  - Cork University Hospital, Cork
  - St James' Hospital, Dublin
  - University Hospital Galway, Galway
  - University Hospital Limerick, Limerick
  - University Hospital Waterford, Waterford

IPD SHARING:
Plan to Share IPD: No